CLINICAL TRIAL: NCT01541215
Title: Efficacy and Safety of Liraglutide in Combination With Metformin Versus Metformin Monotherapy on Glycaemic Control in Children and Adolescents With Type 2 Diabetes
Brief Title: Efficacy and Safety of Liraglutide in Combination With Metformin Compared to Metformin Alone, in Children and Adolescents With Type 2 Diabetes
Acronym: Ellipse™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-3659; 2011-002605-29 (EudraCT Number); P/288/2010 (Other: EMA (PDCO)); U1111-1121-8743 (Other: WHO); CTRI/2013/10/004082 (Registry Identifier: Clinical Trials Registry - India (CTRI))
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lira + Met (Experimental)
  Interventions: Drug: liraglutide; Drug: metformin
- Placebo + Met (Placebo Comparator)
  Interventions: Drug: placebo; Drug: metformin

INTERVENTIONS:
Drug: liraglutide — Administered subcutaneously (s.c., under the skin) once daily.1.8 mg or maximum tolerated dose (MTD: 0.6 mg, 1.2 mg, 1.8 mg) for 26 weeks. Subjects will continue treatment in a 26 week open-labelled extension. Rescue treatment will be allowed if rescue criteria are met.
  Arms: Lira + Met
Drug: placebo — Administered subcutaneously (s.c., under the skin) once daily for 26 weeks. Subjects will discontinue placebo treatment in the open-labelled extension. Rescue treatment will be allowed if rescue criteria are met.
  Arms: Placebo + Met
Drug: metformin — Tablets administered for 26 weeks. Maximum tolerated dose (MTD) between 1000-2000 mg at the discretion of the investigator. Subjects will continue treatment in a 26 week open-labelled extension.

SUMMARY:
This trial is conducted globally. The aim of this trial is to assess the efficacy and safety of liraglutide in the paediatric population in order to potentially address the unmet need for treatment of children and adolescents with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria: - Children and adolescents between the ages of 10-16 years. Subjects cannot turn 17 years and 11 months before the end of treatment (52 weeks) - Diagnosis of type 2 diabetes mellitus and treated for at least 30 days with: diet and exercise alone, diet and exercise in combination with metformin monotherapy, diet and exercise in combination with metformin and a stable (Stable is defined as basal insulin adjustments up to 15%) dose of basal insulin, diet and exercise in combination with a stable (Stable is defined as basal insulin adjustments up to 15%) dose of basal insulin - HbA1c: 7.0-11% (inclusive) if diet and exercise treated or 6.5-11% (inclusive) if treated with metformin as monotherapy, basal insulin as monotherapy or metformin and basal insulin in combination - Body mass index (BMI) above 85% percentile of the general age and gender matched population Exclusion Criteria: - Type 1 diabetes - Maturity onset diabetes of the young (MODY) - Use of any antidiabetic agent other than metformin and/or basal insulin within 90 days prior to screening - Recurrent severe hypoglycaemia or hypoglycaemic unawareness as judged by the investigator - History of chronic pancreatitis or idiopathic acute pancreatitis - Any clinically significant disorder, except for conditions associated with type 2 diabetes history which in the investigator's opinion could interfere with results of the trial - Uncontrolled hypertension, treated or untreated above 99th percentile for age and gender in children - Known or suspected abuse of alcohol or drugs/narcotics

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2012-11-13 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (158):
- United States (60):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Corona, California
  - Novo Nordisk Investigational Site, Costa Mesa, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Moreno Valley, California
  - Novo Nordisk Investigational Site, Palo Alto, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, New Haven, Connecticut
  - Novo Nordisk Investigational Site, Wilmington, Delaware
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Columbus, Georgia
  - Novo Nordisk Investigational Site, Bloomington, Indiana
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Silver Spring, Maryland
  - Novo Nordisk Investigational Site, Worcester, Massachusetts
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Grand Rapids, Michigan
  - Novo Nordisk Investigational Site, Saint Paul, Minnesota
  - Novo Nordisk Investigational Site, Columbia, Missouri
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Hackensack, New Jersey
  - Novo Nordisk Investigational Site, West Orange, New Jersey
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Sleepy Hollow, New York
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Greenville, South Carolina
  - Novo Nordisk Investigational Site, Rapid City, South Dakota
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Edinburg, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Kerrville, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Charlottesville, Virginia
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Charleston, West Virginia
- Novo Nordisk Investigational Site, Ipswich, Queensland, Australia
- Austria (4):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Innsbruck
  - Novo Nordisk Investigational Site, Salzburg
  - Novo Nordisk Investigational Site, Wels
- Belgium (2):
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Leuven
- Novo Nordisk Investigational Site, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (4):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, Westmount, Quebec
- Croatia (2):
  - Novo Nordisk Investigational Site, Rijeka
  - Novo Nordisk Investigational Site, Zagreb
- Denmark (2):
  - Novo Nordisk Investigational Site, Herlev
  - Novo Nordisk Investigational Site, Næstved
- Egypt (3):
  - Novo Nordisk Investigational Site, Al Mansurah
  - Novo Nordisk Investigational Site, Alexandria
  - Novo Nordisk Investigational Site, Cairo
- France (2):
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Montpellier
- Germany (2):
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Mayen
- Greece (3):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Goudi/ Athens
  - Novo Nordisk Investigational Site, Thessaloniki
- Hungary (3):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Miskolc
  - Novo Nordisk Investigational Site, Szombathely
- India (13):
  - Novo Nordisk Investigational Site, Guntur, Andhra Pradesh
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Chandigarh, Punjab
  - Novo Nordisk Investigational Site, Ludhiana, Punjab
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Hyderbad, Telangana
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Kolkata
- Israel (5):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Novo Nordisk Investigational Site, Roma, Italy
- Lebanon (2):
  - Novo Nordisk Investigational Site, Hazmiyeh
  - Novo Nordisk Investigational Site, Lebanon - Beirut
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Mexico (2):
  - Novo Nordisk Investigational Site, Tampico, Tamaulipas
  - Novo Nordisk Investigational Site, Puebla City
- Morocco (2):
  - Novo Nordisk Investigational Site, Fes
  - Novo Nordisk Investigational Site, Rabat
- Novo Nordisk Investigational Site, 's-Hertogenbosch, Netherlands
- Novo Nordisk Investigational Site, Grafton, New Zealand
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Novo Nordisk Investigational Site, Bergen, Norway
- Poland (3):
  - Novo Nordisk Investigational Site, Katowice
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Portugal (2):
  - Novo Nordisk Investigational Site, Braga
  - Novo Nordisk Investigational Site, Lisbon
- Novo Nordisk Investigational Site, Ponce, Puerto Rico
- Romania (3):
  - Novo Nordisk Investigational Site, Timișoara, Timiș County
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Constanța
- Russia (8):
  - Novo Nordisk Investigational Site, Chelyabinsk
  - Novo Nordisk Investigational Site, Izhevsk
  - Novo Nordisk Investigational Site, Krasnoyarsk
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Tomsk
- Serbia (3):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Novi Sad
- Spain (4):
  - Novo Nordisk Investigational Site, Leganés
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Vigo
  - Novo Nordisk Investigational Site, Vitoria-Gasteiz
- Sweden (3):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Huddinge
  - Novo Nordisk Investigational Site, Uppsala
- Taiwan (2):
  - Novo Nordisk Investigational Site, Tainan
  - Novo Nordisk Investigational Site, Taoyuan District
- Thailand (2):
  - Novo Nordisk Investigational Site, Bangkok
  - Novo Nordisk Investigational Site, Chiang Mai
- Turkey (Türkiye) (3):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Kocaeli
- United Kingdom (5):
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Norwich
  - Novo Nordisk Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/sharing-results

REFERENCES:
- [Background] Tamborlane WV, Barrientos-Perez M, Fainberg U, Frimer-Larsen H, Hafez M, Hale PM, Jalaludin MY, Kovarenko M, Libman I, Lynch JL, Rao P, Shehadeh N, Turan S, Weghuber D, Barrett T; Ellipse Trial Investigators. Liraglutide in Children and Adolescents with Type 2 Diabetes. N Engl J Med. 2019 Aug 15;381(7):637-646. doi: 10.1056/NEJMoa1903822. Epub 2019 Apr 28. PMID 31034184
- [Derived] Bensignor MO, Bomberg EM, Bramante CT, Divyalasya TVS, Hale PM, Ramesh CK, Rudser KD, Kelly AS. Effect of liraglutide treatment on body mass index and weight parameters in children and adolescents with type 2 diabetes: Post hoc analysis of the ellipse trial. Pediatr Obes. 2021 Aug;16(8):e12778. doi: 10.1111/ijpo.12778. Epub 2021 Feb 25. PMID 33634589
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 84 sites in 25 countries.
Pre-assignment Details: Eligible subjects entered an 11- to 12-week run-in period where they were to undergo a 3-4 week titration of metformin to a maximum tolerated dose of metformin (≥1000 mg and ≤2000 mg per day) followed by an 8-week maintenance period.
Groups:
- Liraglutide 1.8 mg: After the run-in period, subjects were randomized to receive liraglutide subcutaneous injections once daily (in combination with metformin with or without basal insulin, on a background of diet and exercise) for 52 weeks (26 weeks double blind treatment period followed by a 26-week open-label extension period). The liraglutide dosing was started at 0.6 mg/day during the first week and escalated in weekly increments of 0.6 mg over the following 2-3 weeks. Dose escalation was based on tolerability, as judged by the investigator and on the average of three fasting plasma glucose (FPG) measurements performed by the subject at home on the 3 consecutive days before the dose escalation visit being >6.1 mmol/L (110 mg/dL). Subjects were treated with doses of 0.6, 1.2 or 1.8 after dose escalation. Subjects treated with liraglutide for more than 3 months were asked to return for follow-up visits one and two years after the end of the open label period (after trial drug cessation at week 52).
- Placebo: After the run-in period, subjects were randomized to receive placebo (in combination with metformin with or without basal insulin, on a background of diet and exercise) for a 26 weeks double blind treatment period. The liraglutide placebo was administered once daily subcutaneously in equivalent volume as liraglutide. After 26 weeks, participants discontinued placebo and continued treatment with metformin (with or without basal insulin) during the open-label period.
Period: Treatment Period (52 Weeks)
Arm/Group | Liraglutide 1.8 mg | Placebo
Started | 66 | 69
Exposed | 66 | 68
Completed | 56 | 53
Not Completed | 10 | 16
Not completed — Withdrawal criteria | 6 | 8
Not completed — Non-compliance | 4 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Unclassified | 0 | 3
Period: Follow up 1 (Weeks 53-104)
Arm/Group | Liraglutide 1.8 mg | Placebo
Started | 52 (Subjects who attended safety follow up visit at week 104 were included.) | 0 (Follow up was not planned for the subjects who received placebo.)
Completed | 50 | 0
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Follow up 2 (Weeks 105-156)
Arm/Group | Liraglutide 1.8 mg | Placebo
Started | 48 (Subjects who attended safety follow up visit at week 156 were included.) | 0
Completed | 48 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) - included all randomised subjects receiving at least one dose of liraglutide/placebo
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide 1.8 mg | Placebo | Total
Number analyzed (Participants) | 66 | 68 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.57 (1.73) | 14.57 (1.73) | 14.57 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 83
  Male | 25 | 26 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 23 | 39
  Not Hispanic or Latino | 50 | 45 | 95
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 10 | 8 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 42 | 45 | 87
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 7 | 10
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 7.87 (1.35) | 7.69 (1.34) | 7.78 (1.34)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin)
Description: Change in HbA1c from baseline to week 26. All available data were used for the primary analysis, including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 66 | 68
Percentage of HbA1c | -0.643 (0.215) | 0.415 (0.216)
Statistical Analysis 1: Comparison: Liraglutide 1.8 mg vs Placebo; Analysis using a pattern mixture model of observed data with missing observations imputed from the placebo arm based on multiple (x10.000) imputations. The data for week 26 were then analysed with an ANCOVA model containing treatment, sex and age group as fixed effects and baseline value as covariate. The estimated treatment differences and confidence intervals were combined using Rubins formula; Test type: Superiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 1: Primary analysis: change from baseline to week 26 in HbA1c Superiority of liraglutide over placebo was to be concluded if the 95% confidence interval for the treatment difference for change from baseline in HbA1c (%) after 26 weeks of randomised treatment was entirely below 0%, implying that the two sided p-value was less than 5%; p < 0.001, Pattern Mixture Model; Treatment difference = -1.058, 95% CI 2-sided [-1.653 to -0.464], Standard Error of Mean 0.304

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change in FPG from baseline to week 26. All available data were used for the analysis, including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 66 | 68
mmol/L | -1.076 (0.436) | 0.801 (0.449)
Statistical Analysis 1: Comparison: Liraglutide 1.8 mg vs Placebo; Analysis using a pattern mixture model of observed data with missing observations imputed from the placebo arm based on multiple (x10.000) imputations. The data for weeks 26 were then analysed with an ANCOVA model containing treatment, sex and age group as fixed effects and baseline value as covariate. The estimated treatment differences and confidence intervals were combined using Rubins formula; Test type: Superiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 2: Change from baseline in FPG after 26 weeks of treatment; p = 0.002, Pattern Mixture Model; Treatment difference = -1.878, 95% CI 2-sided [-3.093 to -0.662], Standard Error of Mean 0.620

3. Secondary Outcome: Number of Subjects Having HbA1c Below 7.0%
Description: Percentage of subjects having HbA1c <7.0%. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 26
Population: Full analysis set.
Measure: Number; unit: Percentage of subjects
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 66 | 68
Percentage of subjects | 63.7 | 36.5
Statistical Analysis 1: Comparison: Liraglutide 1.8 mg vs Placebo; Missing data was imputed using pattern mixture model. For each imputed data set the binary response was analysed in a logistic regression model using a logit link with treatment and stratification group (gender*age group) as fixed factors and baseline HbA1c as covariate.The estimated treatment effects and confidence intervals were combined using Rubin´s formula; Test type: Superiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 3: HbA1c < 7.0% after 26 weeks of treatment; p < 0.001, logistic regression model; Treatment odds ratio = 5.353, 95% CI 2-sided [2.105 to 13.615]

4. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) Standard Deviation Score (SDS)
Description: Change in BMI SDS from baseline to week 26. BMI SDS was calculated using the following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' BMI provided for each sex and age. For each subject, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The method is described in the world health organisation (WHO) Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set.
Measure: Least Squares Mean (Standard Error); unit: SDS score
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 66 | 68
SDS score | -0.254 (0.039) | -0.208 (0.039)
Statistical Analysis 1: Comparison: Liraglutide 1.8 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 4: Change from baseline in BMI SDS after 26 weeks of treatment; p = 0.392, Pattern Mixture Model; Treatment difference = -0.047, 95% CI 2-sided [-0.153 to 0.060], Standard Error of Mean 0.055

5. Secondary Outcome: Number of Subjects Having HbA1c Below 7.0%
Description: Number of subjects achieving HbA1c <7.0% after 52 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 52
Participants
  Yes | 27 | 16
  No | 29 | 36

6. Secondary Outcome: Number of Subjects Having HbA1c Maximum 6.5%
Description: Number of subjects achieving HbA1c <=6.5% after 26 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 59 | 58
Participants
  Yes | 28 | 19
  No | 31 | 39

7. Secondary Outcome: Number of Subjects Having HbA1c Maximum 6.5%
Description: Number of subjects achieving HbA1c <=6.5% after 52 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 52
Participants
  Yes | 25 | 13
  No | 31 | 39

8. Secondary Outcome: Number of Subjects Having HbA1c Below 7.0% Without Severe or Minor Hypoglycaemic Episodes
Description: Number of subjects achieving HbA1c <7.0% without severe or minor hypoglycaemic episodes after 26 weeks.
  Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
  Minor hypoglycaemia was defined as meeting either of the below criteria:
  1. an episode with symptoms consistent with hypoglycaemia with confirmation by blood glucose <2.8 mmol/L (50 mg/dL) or plasma glucose <3.1 mmol/L (56 mg/dL), and which was handled by the subject him/herself
  2. any asymptomatic blood glucose value <2.8 mmol/L (50 mg/dL) or plasma glucose value <3.1 mmol/L (56 mg/dL) All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 59 | 58
Participants
  Yes | 31 | 21
  No | 28 | 37

9. Secondary Outcome: Number of Subjects Having HbA1c Below 7.0% Without Severe or Minor Hypoglycaemic Episodes
Description: Number of subjects achieving HbA1c <7.0% without severe or minor hypoglycaemic episodes after 52 weeks.
  Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
  Minor hypoglycaemia was defined as meeting either of the below criteria:
  1. an episode with symptoms consistent with hypoglycaemia with confirmation by blood glucose <2.8 mmol/L (50 mg/dL) or plasma glucose <3.1 mmol/L (56 mg/dL), and which was handled by the subject him/herself
  2. any asymptomatic blood glucose value <2.8 mmol/L (50 mg/dL) or plasma glucose value <3.1 mmol/L (56 mg/dL) All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 52
Participants
  Yes | 22 | 16
  No | 34 | 36

10. Secondary Outcome: Number of Subjects Having HbA1c Below 7.5%
Description: Number of subjects achieving HbA1c <7.5% after 26 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 59 | 58
Participants
  Yes | 43 | 29
  No | 16 | 29

11. Secondary Outcome: Number of Subjects Having HbA1c Below 7.5%
Description: Number of subjects achieving HbA1c <7.5% after 52 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 52
Participants
  Yes | 36 | 23
  No | 20 | 29

12. Secondary Outcome: Change in HbA1c
Description: Change in HbA1c from baseline to week 52. All available data were used for the analysis, including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 52
percentage of HbA1c | -0.732 (1.423) | 0.677 (1.523)

13. Secondary Outcome: Change in FPG
Description: Change in FPG from baseline to week 52. All available data were used for the analysis, including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 53
mmol/L | -1.627 (2.717) | 0.983 (3.954)

14. Secondary Outcome: Change in Mean 7-point Self-measured Plasma Glucose
Description: Change in mean 7-point self-measured plasma glucose after 26 weeks. Subjects were instructed to measure their plasma glucose at following timepoints: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner and at bedtime. Mean 7-point SMPG was defined as the area under the profile (calculated using the trapezoidal method) divided by time. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 39 | 46
mmol/L | -2.384 (2.638) | 0.198 (2.056)

15. Secondary Outcome: Change From Baseline in 7-point Self-measured Plasma Glucose
Description: Change in mean 7-point self-measured plasma glucose after 52 weeks. Subjects were instructed to measure their plasma glucose at following timepoints: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner and at bedtime. Mean 7-point SMPG was defined as the area under the profile (calculated using the trapezoidal method) divided by time. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 41 | 39
mmol/L | -2.309 (2.968) | -0.748 (1.944)

16. Secondary Outcome: Change in Post-prandial Increments (From Before Meal to 90 Min After Breakfast, Lunch, and Dinner)
Description: Change in post-prandial increments (from before meal to 90 min after breakfast, lunch, and dinner) after 26 weeks. Post-prandial increment for each meal (breakfast, lunch, and dinner) was derived from the 7-point SMPG profile as the difference between post-prandial plasma glucose values and the plasma glucose values before the meal. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of analysed=participants with available data for specified timepoints.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 41 | 46
mmol/L
  Breakfast: number analyzed (Participants) | 37 | 46
  Breakfast | -1.528 (3.168) | -0.319 (3.228)
  Lunch: number analyzed (Participants) | 41 | 43
  Lunch | -0.358 (3.281) | -0.658 (3.421)
  Dinner: number analyzed (Participants) | 38 | 42
  Dinner | 0.397 (3.790) | -0.226 (2.806)

17. Secondary Outcome: Change in Post-prandial Increments (From Before Meal to 90 Min After Breakfast, Lunch, and Dinner)
Description: Change in post-prandial increments (from before meal to 90 min after breakfast, lunch, and dinner) after 52 weeks. Post-prandial increment for each meal (breakfast, lunch, and dinner) was derived from the 7-point SMPG profile as the difference between post-prandial plasma glucose values and the plasma glucose values before the meal. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of analysed=participants with available data for specified timepoints.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 42 | 38
mmol/L
  Breakfast | -1.802 (3.338) | 0.053 (2.124)
  Lunch: number analyzed (Participants) | 42 | 36
  Lunch | -0.735 (3.809) | -1.219 (3.038)
  Dinner: number analyzed (Participants) | 38 | 36
  Dinner | -0.028 (3.501) | -0.195 (2.803)

18. Secondary Outcome: Change in Mean Post-prandial Increment Across All Three Meals (Breakfast, Lunch, and Dinner)
Description: Change in mean post-prandial increment across all three meals (breakfast, lunch, and dinner) after 26 weeks. Post-prandial increment for each meal (breakfast, lunch, and dinner) was derived from the 7-point SMPG profile as the difference between post-prandial plasma glucose values and the plasma glucose values before the meal. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 40 | 46
mmol/L | -0.428 (2.172) | -0.362 (1.733)

19. Secondary Outcome: Change in Mean Post-prandial Increment Across All Three Meals (Breakfast, Lunch, and Dinner)
Description: Change in mean post-prandial increment across all three meals (breakfast, lunch, and dinner) after 52 weeks. Post-prandial increment for each meal (breakfast, lunch, and dinner) was derived from the 7-point SMPG profile as the difference between post-prandial plasma glucose values and the plasma glucose values before the meal. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 41 | 39
mmol/L | -0.747 (2.245) | -0.397 (1.594)

20. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight after 26 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 60 | 58
kg | -2.48 (5.59) | -0.87 (3.84)

21. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight after 52 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 53
kg | -2.27 (8.05) | 1.02 (4.64)

22. Secondary Outcome: Change From Baseline in BMI Standard Deviation Score (SDS)
Description: Change in BMI SDS from baseline to week 52. BMI SDS was calculated using the following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' BMI provided for each sex and age. For each subject, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The method is described in the WHO Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: SDS score
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 53
SDS score | -0.361 (0.542) | -0.166 (0.330)

23. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic Blood Pressure)
Description: Change in blood pressure (systolic and diastolic blood pressure) after 26 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 60 | 58
mmHg
  Systolic Blood Pressure | -1.65 (10.69) | 0.03 (10.05)
  Diastolic Blood Pressure | -1.27 (8.39) | 0.97 (7.65)

24. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic Blood Pressure)
Description: Change in blood pressure (systolic and diastolic blood pressure) after 52 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 53
mmHg
  Systolic Blood Pressure | -0.77 (11.77) | 2.81 (8.48)
  Diastolic Blood Pressure | 0.46 (10.01) | 1.83 (7.26)

25. Secondary Outcome: Ratio to Baseline: Fasting Insulin
Description: Ratio to baseline (fasting insulin) at week 26. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 59 | 57
ratio | 0.9 (76.4) | 1.0 (77.9)

26. Secondary Outcome: Ratio to Baseline: Fasting Insulin
Description: Ratio to baseline (fasting insulin) at week 52. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 54 | 53
ratio | 1.0 (80.6) | 1.1 (142.8)

27. Secondary Outcome: Ratio to Baseline: Fasting Pro-insulin
Description: Ratio to baseline (fasting pro-insulin) at week 26. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 55
ratio | 0.62 (110.3) | 0.88 (131.6)

28. Secondary Outcome: Ratio to Baseline: Fasting Pro-insulin
Description: Ratio to baseline (fasting pro-insulin) at week 52. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 54 | 49
ratio | 0.62 (118.0) | 0.79 (121.0)

29. Secondary Outcome: Ratio to Baseline: Pro-insulin/Insulin Ratio
Description: Ratio to baseline (Pro-insulin/insulin ratio) after week 26. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 55 | 54
ratio | 0.690 (102.4) | 0.923 (197.6)

30. Secondary Outcome: Ratio to Baseline: Pro-insulin/Insulin Ratio
Description: Ratio to baseline (Pro-insulin/insulin ratio) after week 52. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 53 | 49
ratio | 0.689 (106.6) | 0.770 (225.1)

31. Secondary Outcome: Ratio to Baseline: Fasting Glucagon
Description: Ratio to baseline (fasting glucagon) at week 26. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 60 | 57
ratio | 0.98 (29.3) | 1.03 (32.4)

32. Secondary Outcome: Ratio to Baseline: Fasting Glucagon
Description: Ratio to baseline (fasting glucagon) at week 52. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 54 | 52
ratio | 1.01 (35.0) | 1.05 (32.7)

33. Secondary Outcome: Ratio to Baseline: Fasting C-peptide
Description: Ratio to baseline (fasting C-peptide) at week 26. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 59 | 58
ratio | 0.93 (39.7) | 0.84 (82.3)

34. Secondary Outcome: Ratio to Baseline: Fasting C-peptide
Description: Ratio to baseline (fasting C-peptide) at week 52. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 54 | 53
ratio | 0.94 (40.8) | 0.83 (56.5)

35. Secondary Outcome: Ratio to Baseline: Homeostasis Model Assessment of Beta-cell Function (HOMA-B)
Description: Ratio to baseline (HOMA-B) after 26 weeks. HOMA-B is an index of beta-cell function and was calculated from fasting insulin. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 51
ratio | 1.24 (96.9) | 1.01 (119.0)

36. Secondary Outcome: Ratio to Baseline: HOMA-B
Description: Ratio to baseline (HOMA-B) after 52 weeks. HOMA-B is an index of beta-cell function and was calculated from fasting insulin. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 51 | 49
ratio | 1.48 (105.0) | 0.93 (166.8)

37. Secondary Outcome: Ratio to Baseline: Homeostasis Model Assessment as an Index of Insulin Resistance (HOMA-IR)
Description: Ratio to baseline (HOMA-IR) after 26 weeks. HOMA-IR is an index of insulin resistance and was calculated from fasting insulin. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 58 | 54
ratio | 0.73 (80.5) | 0.98 (80.8)

38. Secondary Outcome: Ratio to Baseline: HOMA-IR
Description: Ratio to baseline (HOMA-IR) after 52 weeks. HOMA-IR is an index of insulin resistance and was calculated from fasting insulin. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 53 | 52
ratio | 0.82 (86.4) | 1.08 (140.3)

39. Secondary Outcome: Ratio to Baseline: Total Cholesterol
Description: Ratio to baseline (total cholesterol) after 26 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 60 | 58
ratio | 0.975 (17.7) | 1.008 (13.3)

40. Secondary Outcome: Ratio to Baseline: Total Cholesterol
Description: Ratio to baseline (total cholesterol) after 52 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 52
ratio | 1.013 (21.0) | 1.026 (13.5)

41. Secondary Outcome: Ratio to Baseline: Low Density Lipoprotein (LDL) Cholesterol
Description: Ratio to baseline (LDL cholesterol) after 26 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 58 | 57
ratio | 0.998 (24.8) | 0.993 (20.4)

42. Secondary Outcome: Ratio to Baseline: LDL Cholesterol
Description: Ratio to baseline (LDL cholesterol) after 52 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 54 | 48
ratio | 1.042 (46.3) | 1.035 (21.5)

43. Secondary Outcome: Ratio to Baseline: Very Low-density Lipoprotein (VLDL) Cholesterol
Description: Ratio to baseline (VLDL cholesterol) after 26 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 59 | 58
ratio | 0.890 (51.6) | 1.035 (35.3)

44. Secondary Outcome: Ratio to Baseline: VLDL Cholesterol
Description: Ratio to baseline (VLDL cholesterol) after 52 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 51
ratio | 0.983 (48.4) | 1.003 (45.5)

45. Secondary Outcome: Ratio to Baseline: High-density Lipoprotein (HDL) Cholesterol
Description: Ratio to baseline (HDL cholesterol) after 26 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 59 | 58
ratio | 0.997 (18.7) | 0.981 (16.3)

46. Secondary Outcome: Ratio to Baseline: HDL Cholesterol
Description: Ratio to baseline (HDL cholesterol) after 52 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 51
ratio | 1.028 (16.0) | 1.000 (18.8)

47. Secondary Outcome: Ratio to Baseline: Triglycerides
Description: Ratio to baseline (triglycerides) after 26 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 60 | 58
ratio | 0.894 (50.6) | 1.038 (36.0)

48. Secondary Outcome: Ratio to Baseline: Triglycerides
Description: Ratio to baseline (triglycerides) after 52 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 53
ratio | 0.964 (50.5) | 1.036 (48.4)

49. Secondary Outcome: Ratio to Baseline: Free Fatty Acids
Description: Ratio to baseline (free fatty acids) after 26 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 59 | 58
ratio | 1.023 (67.4) | 0.985 (47.5)

50. Secondary Outcome: Ratio to Baseline: Free Fatty Acids
Description: Ratio to baseline (free fatty acids) after 52 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of participants analysed=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 54 | 51
ratio | 0.928 (58.2) | 0.868 (54.8)

51. Secondary Outcome: Change From Baseline in Pulse
Description: Change from baseline in pulse 26 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Safety analysis set - included all subjects receiving at least one dose of liraglutide/placebo (134 subjects). Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 60 | 58
beats/minute | 1.40 (10.89) | 0.33 (7.69)

52. Secondary Outcome: Change From Baseline in Pulse
Description: Change from baseline in pulse 52 weeks. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Safety analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 53
beats/minute | -0.05 (10.39) | -0.28 (7.88)

53. Secondary Outcome: Change From Baseline in Height SDS
Description: Change in height SDS from baseline to week 26. Height SDS was calculated using the following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' height provided for each sex and age. For each subject, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The method is described in the WHO Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Safety analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: SDS score
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 60 | 58
SDS score | -0.100 (0.133) | -0.042 (0.210)

54. Secondary Outcome: Change From Baseline in Height SDS
Description: Change in height SDS from baseline to week 52. Height SDS was calculated using the following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' height provided for each sex and age. For each subject, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The method is described in the WHO Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Safety analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: SDS score
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 53
SDS score | -0.192 (0.223) | -0.134 (0.293)

55. Secondary Outcome: Change in Bone Age Assessment (X-ray of Left Hand and Wrist)
Description: Change in bone age from baseline to week 52. If the baseline (week 0) bone age assessment indicated that all epiphyses were fused, then the assessment was not repeated at week 52.
Time Frame: Week 0, week 52
Population: Safety analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 31 | 26
years | 1.197 (0.899) | 1.088 (0.889)

56. Secondary Outcome: Pubertal Assessment/Progression (Tanner Staging)
Description: Pubertal development was assessed in 3 areas (breast, penis and pubic hair development) by the Tanner staging in accordance with stages I-V. The Tanner staging assessment was no longer required to be performed once a subject reached the Tanner stage V, as judged by the investigator. Reported results are number of participants at different Tanner stages at week 0, week 26 and week 52.
Time Frame: Week 0, week 26, week 52
Population: Safety analysis set. Number of participants analysed=participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 66 | 68
Participants
  Female - Breast development - Week 0: number analyzed (Participants) | 41 | 42
  Female - Breast development - Week 0: Stage I | 1 | 0
  Female - Breast development - Week 0: Stage II | 2 | 0
  Female - Breast development - Week 0: Stage III | 4 | 10
  Female - Breast development - Week 0: Stage IV | 8 | 9
  Female - Breast development - Week 0: Stage V | 26 | 23
  Female - Breast development - Week 26: number analyzed (Participants) | 37 | 36
  Female - Breast development - Week 26: Stage I | 0 | 0
  Female - Breast development - Week 26: Stage II | 1 | 0
  Female - Breast development - Week 26: Stage III | 2 | 4
  Female - Breast development - Week 26: Stage IV | 5 | 10
  Female - Breast development - Week 26: Stage V | 29 | 22
  Female - Breast development - Week 52: number analyzed (Participants) | 33 | 33
  Female - Breast development - Week 52: Stage I | 0 | 0
  Female - Breast development - Week 52: Stage II | 0 | 0
  Female - Breast development - Week 52: Stage III | 1 | 2
  Female - Breast development - Week 52: Stage IV | 5 | 9
  Female - Breast development - Week 52: Stage V | 27 | 22
  Male - Penis Development - Week 0: number analyzed (Participants) | 25 | 26
  Male - Penis Development - Week 0: Stage I | 2 | 0
  Male - Penis Development - Week 0: Stage II | 1 | 3
  Male - Penis Development - Week 0: Stage III | 2 | 6
  Male - Penis Development - Week 0: Stage IV | 9 | 11
  Male - Penis Development - Week 0: Stage V | 11 | 6
  Male - Penis Development - Week 26: number analyzed (Participants) | 25 | 23
  Male - Penis Development - Week 26: Stage I | 2 | 0
  Male - Penis Development - Week 26: Stage II | 1 | 1
  Male - Penis Development - Week 26: Stage III | 2 | 4
  Male - Penis Development - Week 26: Stage IV | 7 | 8
  Male - Penis Development - Week 26: Stage V | 13 | 10
  Male - Penis Development - Week 52: number analyzed (Participants) | 25 | 21
  Male - Penis Development - Week 52: Stage I | 1 | 0
  Male - Penis Development - Week 52: Stage II | 2 | 0
  Male - Penis Development - Week 52: Stage III | 0 | 2
  Male - Penis Development - Week 52: Stage IV | 7 | 6
  Male - Penis Development - Week 52: Stage V | 15 | 13
  Pubic Hair Development - Week 0: number analyzed (Participants) | 66 | 67
  Pubic Hair Development - Week 0: Stage I | 3 | 3
  Pubic Hair Development - Week 0: Stage II | 3 | 0
  Pubic Hair Development - Week 0: Stage III | 8 | 10
  Pubic Hair Development - Week 0: Stage IV | 14 | 25
  Pubic Hair Development - Week 0: Stage V | 38 | 29
  Pubic Hair Development - Week 26: number analyzed (Participants) | 62 | 58
  Pubic Hair Development - Week 26: Stage I | 3 | 0
  Pubic Hair Development - Week 26: Stage II | 0 | 2
  Pubic Hair Development - Week 26: Stage III | 5 | 4
  Pubic Hair Development - Week 26: Stage IV | 11 | 18
  Pubic Hair Development - Week 26: Stage V | 43 | 34
  Pubic Hair Development - Week 52: number analyzed (Participants) | 57 | 53
  Pubic Hair Development - Week 52: Stage I | 1 | 0
  Pubic Hair Development - Week 52: Stage II | 1 | 0
  Pubic Hair Development - Week 52: Stage III | 4 | 2
  Pubic Hair Development - Week 52: Stage IV | 8 | 17
  Pubic Hair Development - Week 52: Stage V | 43 | 34

57. Secondary Outcome: Growth (Height Velocity)
Description: Growth (i.e., height velocity) is the change in height per year and is measured in cm/year. The height velocity was calculated as the difference between current height and height at baseline (week 0) divided by the time (in days) between those measurement time points and multiplied by 365 days.
Time Frame: Week 0, week 26
Population: Safety analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 60 | 58
cm/year | 1.633 (2.016) | 2.486 (2.834)

58. Secondary Outcome: Growth (Height Velocity)
Description: as for outcome 57
Time Frame: Week 0, week 52
Population: Safety analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 56 | 53
cm/year | 1.345 (1.730) | 1.817 (2.043)

59. Secondary Outcome: Height Velocity SDS
Description: Height velocity SDS scores at week 26. Height velocity is change in height per year. The height velocity was calculated as the difference between current height and height at baseline (week 0) divided by time between those measurement time points and multiplied by 365 days. Height velocity SDS was calculated using following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' height provided for each sex and age. For each subject, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The method is described in the WHO Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Safety analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: SDS score
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 60 | 58
SDS score | -1.24 (1.695) | -0.557 (2.058)

60. Secondary Outcome: Height Velocity SDS
Description: Height velocity SDS scores at week 52. Height velocity is change in height per year. The height velocity was calculated as the difference between current height and height at baseline (week 0) divided by time between those measurement time points and multiplied by 365 days. Height velocity SDS was calculated using following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' height provided for each sex and age. For each subject, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The method is described in the WHO Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Safety analysis set. Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: SDS score
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 52 | 48
SDS score | -0.887 (1.460) | -0.551 (1.711)

61. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: Total number of hypoglycaemic episodes according to American Diabetes Association (ADA) classification from baseline (week 0) to week 26.
Time Frame: 0-26 weeks
Population: Safety analysis set
Measure: Number; unit: hypoglycaemic episodes
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 66 | 68
hypoglycaemic episodes | 92 | 43

62. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: Total number of hypoglycaemic episodes according to American Diabetes Association (ADA) classification from baseline (week 0) to week 52.
Time Frame: 0-52 weeks
Population: Safety analysis set
Measure: Number; unit: hypoglycaemic episodes
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 66 | 68
hypoglycaemic episodes | 160 | 63

63. Secondary Outcome: Number of Adverse Events (Week 0-26)
Description: Total number of adverse events during 26 weeks.
Time Frame: 0-26 weeks
Population: Safety analysis set
Measure: Number; unit: events
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 66 | 68
events | 310 | 230

64. Secondary Outcome: Number of Adverse Events (Week 0-52)
Description: Total number of adverse events during entire treatment period.
Time Frame: 0-52 weeks
Population: Safety analysis set
Measure: Number; unit: events
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 66 | 68
events | 426 | 321

65. Secondary Outcome: Number of Serious Adverse Events (Week 0-26)
Description: Total number of serious adverse events during 26 weeks.
Time Frame: 0-26 weeks
Population: Safety analysis set
Measure: Number; unit: events
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 66 | 68
events | 7 | 4

66. Secondary Outcome: Number of Serious Adverse Events (Week 0-52)
Description: Total number of serious adverse events during entire treatment period.
Time Frame: 0-52 weeks
Population: Safety analysis set
Measure: Number; unit: events
Arm/Group | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 66 | 68
events | 10 | 5

67. Secondary Outcome: Number of Adverse Events (Week 53-104)
Description: This outcome is applicable only for the Liraglutide 1.8 mg treatment arm. Number of adverse events reported during follow-up 1 (week 53 to 104).
Time Frame: Week 53-104
Population: Safety analysis set- Subjects who received liraglutide for more than 3 months during the treatment period (week 0-52) and provided safety follow-up data anytime during week 53-104.
Measure: Number; unit: events
Groups:
- Liraglutide 1.8 mg: Follow-up 1: Subjects who received liraglutide for more than 3 months during the treatment period (week 0-52), were followed-up at week 104.
Arm/Group | Liraglutide 1.8 mg: Follow-up 1
Number analyzed (Participants) | 52
events | 30

68. Secondary Outcome: Number of Serious Adverse Events (Week 53-104)
Description: This outcome is applicable only for the Liraglutide 1.8 mg treatment arm. Number of serious adverse events reported during follow up 1 (week 53 to 104).
Time Frame: Weeks 53-104
Population: as for outcome 67
Measure: Number; unit: events
Arm/Group | Liraglutide 1.8 mg: Follow-up 1
Number analyzed (Participants) | 52
events | 7

69. Secondary Outcome: Growth (Height Velocity)- Week 104
Description: Growth (i.e., height velocity) is the change in height per year and is measured in cm/year. The height velocity was calculated as the difference between current height and height at baseline (week 0) divided by the time (in days) between those measurement time points and multiplied by 365 days. This outcome is applicable only for the Liraglutide 1.8 mg treatment arm.
Time Frame: Week 0, week 104
Population: Safety analysis set- Subjects who received liraglutide for more than 3 months during the treatment period (week 0-52) and provided safety follow-up data anytime during week 53-104. Overall number of participants analyzed= subjects with available data.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Liraglutide 1.8 mg: Follow-up 1
Number analyzed (Participants) | 50
cm/year | 1.149 (1.776)

70. Secondary Outcome: Height Velocity SDS- Week 104
Description: The height velocity was calculated as the difference between current height and height at baseline (week 0) divided by time between those measurement time points and multiplied by 365 days. Height velocity SDS was calculated using following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' height provided for each sex and age. For each subject, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The method is described in the WHO Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. This outcome is applicable only for the Liraglutide 1.8 mg treatment arm.
Time Frame: Week 0, week 104
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: SDS score
Arm/Group | Liraglutide 1.8 mg: Follow-up 1
Number analyzed (Participants) | 41
SDS score | -0.523 (1.466)

71. Secondary Outcome: Change From Week 52 in Height SDS- Week 104
Description: Change in height SDS from week 52 to week 104. Height SDS was calculated using the following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' height provided for each sex and age. For each subject, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The method is described in the WHO Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication. This outcome is applicable only for the Liraglutide 1.8 mg treatment arm.
Time Frame: Week 52, week 104
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: SDS score
Arm/Group | Liraglutide 1.8 mg: Follow-up 1
Number analyzed (Participants) | 49
SDS score | -0.133 (0.338)

72. Secondary Outcome: Change in Pubertal Assessment/Progression (Tanner Staging)- Week 104
Description: Pubertal development was assessed in 3 areas (breast, penis and pubic hair development) by the Tanner staging in accordance with stages I-V, where stage I represents "pre-adoloscent development" and stage V represents "pubertal development equivalent to that of an adult". The Tanner staging assessment was no longer required to be performed once a subject reached the Tanner stage V, as judged by the investigator. Reported results are number of subjects at different Tanner stages at week 52 and week 104. This outcome is applicable only for the Liraglutide 1.8 mg treatment arm.
Time Frame: Week 52, week 104
Population: Safety analysis set- Subjects who received liraglutide for more than 3 months during the treatment period (week 0-52) and provided safety follow-up data anytime during week 53-104. Number analyzed= subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg: Follow-up 1
Number analyzed (Participants) | 52
Participants
  Female- Breast development- Week 52: number analyzed (Participants) | 27
  Female- Breast development- Week 52: Stage I | 0
  Female- Breast development- Week 52: Stage II | 0
  Female- Breast development- Week 52: Stage III | 1
  Female- Breast development- Week 52: Stage IV | 5
  Female- Breast development- Week 52: Stage V | 21
  Female- Breast development- Week 104: number analyzed (Participants) | 16
  Female- Breast development- Week 104: Stage I | 0
  Female- Breast development- Week 104: Stage II | 0
  Female- Breast development- Week 104: Stage III | 0
  Female- Breast development- Week 104: Stage IV | 5
  Female- Breast development- Week 104: Stage V | 11
  Male- Penis development- Week 52: number analyzed (Participants) | 24
  Male- Penis development- Week 52: Stage I | 1
  Male- Penis development- Week 52: Stage II | 2
  Male- Penis development- Week 52: Stage III | 0
  Male- Penis development- Week 52: Stage IV | 7
  Male- Penis development- Week 52: Stage V | 14
  Male- Penis development- Week 104: number analyzed (Participants) | 14
  Male- Penis development- Week 104: Stage I | 0
  Male- Penis development- Week 104: Stage II | 1
  Male- Penis development- Week 104: Stage III | 0
  Male- Penis development- Week 104: Stage IV | 5
  Male- Penis development- Week 104: Stage V | 8
  Female- Pubic hair development- Week 52: number analyzed (Participants) | 26
  Female- Pubic hair development- Week 52: Stage I | 0
  Female- Pubic hair development- Week 52: Stage II | 0
  Female- Pubic hair development- Week 52: Stage III | 2
  Female- Pubic hair development- Week 52: Stage IV | 2
  Female- Pubic hair development- Week 52: Stage V | 22
  Female- Pubic hair development- Week 104: number analyzed (Participants) | 16
  Female- Pubic hair development- Week 104: Stage I | 0
  Female- Pubic hair development- Week 104: Stage II | 0
  Female- Pubic hair development- Week 104: Stage III | 1
  Female- Pubic hair development- Week 104: Stage IV | 2
  Female- Pubic hair development- Week 104: Stage V | 13
  Male- Pubic hair development- Week 52: number analyzed (Participants) | 24
  Male- Pubic hair development- Week 52: Stage I | 1
  Male- Pubic hair development- Week 52: Stage II | 1
  Male- Pubic hair development- Week 52: Stage III | 2
  Male- Pubic hair development- Week 52: Stage IV | 6
  Male- Pubic hair development- Week 52: Stage V | 14
  Male- Pubic hair development- Week 104: number analyzed (Participants) | 14
  Male- Pubic hair development- Week 104: Stage I | 0
  Male- Pubic hair development- Week 104: Stage II | 1
  Male- Pubic hair development- Week 104: Stage III | 0
  Male- Pubic hair development- Week 104: Stage IV | 4
  Male- Pubic hair development- Week 104: Stage V | 9

73. Secondary Outcome: Change From Week 52 in Bone Age Assessment (X-ray of Left Hand and Wrist)- Week 104
Description: Change in bone age from week 52 to week 104. This outcome is applicable only for the Liraglutide 1.8 mg treatment arm.
Time Frame: Week 52, week 104
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Liraglutide 1.8 mg: Follow-up 1
Number analyzed (Participants) | 13
Years | 1.231 (0.992)

74. Secondary Outcome: Number of Adverse Events (Week 53-156)
Description: This outcome measure is applicable only for the Liraglutide 1.8 mg treatment arm. Number of adverse events reported during the follow-up period (weeks 53 to 156).
Time Frame: Week 53-156
Population: Safety analysis set- Subjects who received liraglutide for more than 3 months during the treatment period (week 0-52) and provided safety follow-up data anytime during weeks 53-156.
Measure: Number; unit: events
Groups:
- Liraglutide 1.8 mg: Follow-up 1 and 2: Subjects who received liraglutide for more than 3 months during the treatment period (week 0-52), were followed-up at weeks 104 and 156.
Arm/Group | Liraglutide 1.8 mg: Follow-up 1 and 2
Number analyzed (Participants) | 52
events | 47

75. Secondary Outcome: Number of Serious Adverse Events (Week 53-156)
Description: This outcome measure is applicable only for the Liraglutide 1.8 mg treatment arm. Number of serious adverse events reported during the follow up period (week 53 to 156).
Time Frame: Weeks 53-156
Population: as for outcome 74
Measure: Number; unit: events
Arm/Group | Liraglutide 1.8 mg: Follow-up 1 and 2
Number analyzed (Participants) | 52
events | 9

76. Secondary Outcome: Growth (Height Velocity)- Week 156
Description: Growth (i.e., height velocity) is the change in height per year and is measured in cm/year. The height velocity was calculated as the difference between current height and height at baseline (week 0) divided by the time (in days) between those measurement time points and multiplied by 365 days. This outcome measure is applicable only for the Liraglutide 1.8 mg treatment arm.
Time Frame: Week 0, week 156
Population: Safety analysis set- Subjects who received liraglutide for more than 3 months during the treatment period (week 0-52) and provided safety follow-up data anytime during week 53-156. Overall number of participants analyzed= subjects with available data at week 156.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Liraglutide 1.8 mg: Follow-up 1 and 2
Number analyzed (Participants) | 45
cm/year | 1.100 (1.504)

77. Secondary Outcome: Height Velocity SDS- Week 156
Description: The height velocity was calculated as the difference between current height and height at baseline (week 0) divided by time between those measurement time points and multiplied by 365 days. Height velocity SDS was calculated using following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' height provided for each sex and age. For each subject, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The method is described in the WHO Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. This outcome measure is applicable only for the Liraglutide 1.8 mg treatment arm.
Time Frame: Week 0, week 156
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: SDS score
Arm/Group | Liraglutide 1.8 mg: Follow-up 1 and 2
Number analyzed (Participants) | 27
SDS score | 0.142 (1.156)

78. Secondary Outcome: Change From Week 52 in Height SDS- Week 156
Description: Change in height SDS from week 52 to week 156. Height SDS was calculated using the following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' height provided for each sex and age. For each subject, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The method is described in the WHO Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. All available data were used for the analysis including data collected after treatment discontinuation and initiation of rescue medication. This outcome measure is applicable only for the Liraglutide 1.8 mg treatment arm.
Time Frame: Week 52, week 156
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: SDS score
Arm/Group | Liraglutide 1.8 mg: Follow-up 1 and 2
Number analyzed (Participants) | 36
SDS score | -0.224 (0.446)

79. Secondary Outcome: Change in Pubertal Assessment/Progression (Tanner Staging)- Week 156
Description: Pubertal development was assessed in 3 areas (breast, penis and pubic hair development) by the Tanner staging in accordance with stages I-V, where stage I represents "pre-adoloscent development" and stage V represents "pubertal development equivalent to that of an adult". The Tanner staging assessment was no longer required to be performed once a subject reached the Tanner stage V, as judged by the investigator. Reported results are number of subjects at different Tanner stages at week 52 and week 156. This outcome measure is applicable only for the Liraglutide 1.8 mg treatment arm.
Time Frame: Week 52, week 156
Population: Safety analysis set- Subjects who received liraglutide for more than 3 months during the treatment period (week 0-52) and provided safety follow-up data anytime during week 53-156. Number analyzed= subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg: Follow-up 1 and 2
Number analyzed (Participants) | 52
Participants
  Female- Breast development- Week 52: number analyzed (Participants) | 27
  Female- Breast development- Week 52: Stage I | 0
  Female- Breast development- Week 52: Stage II | 0
  Female- Breast development- Week 52: Stage III | 1
  Female- Breast development- Week 52: Stage IV | 5
  Female- Breast development- Week 52: Stage V | 21
  Female- Breast development- Week 156: number analyzed (Participants) | 14
  Female- Breast development- Week 156: Stage I | 0
  Female- Breast development- Week 156: Stage II | 0
  Female- Breast development- Week 156: Stage III | 0
  Female- Breast development- Week 156: Stage IV | 3
  Female- Breast development- Week 156: Stage V | 11
  Male- Penis development- Week 52: number analyzed (Participants) | 24
  Male- Penis development- Week 52: Stage I | 1
  Male- Penis development- Week 52: Stage II | 2
  Male- Penis development- Week 52: Stage III | 0
  Male- Penis development- Week 52: Stage IV | 7
  Male- Penis development- Week 52: Stage V | 14
  Male- Penis development- Week 156: number analyzed (Participants) | 13
  Male- Penis development- Week 156: Stage I | 0
  Male- Penis development- Week 156: Stage II | 0
  Male- Penis development- Week 156: Stage III | 1
  Male- Penis development- Week 156: Stage IV | 3
  Male- Penis development- Week 156: Stage V | 9
  Female- Pubic hair development- Week 52: number analyzed (Participants) | 26
  Female- Pubic hair development- Week 52: Stage I | 0
  Female- Pubic hair development- Week 52: Stage II | 0
  Female- Pubic hair development- Week 52: Stage III | 2
  Female- Pubic hair development- Week 52: Stage IV | 2
  Female- Pubic hair development- Week 52: Stage V | 22
  Female- Pubic hair development- Week 156: number analyzed (Participants) | 13
  Female- Pubic hair development- Week 156: Stage I | 0
  Female- Pubic hair development- Week 156: Stage II | 0
  Female- Pubic hair development- Week 156: Stage III | 0
  Female- Pubic hair development- Week 156: Stage IV | 2
  Female- Pubic hair development- Week 156: Stage V | 11
  Male- Pubic hair development- Week 52: number analyzed (Participants) | 24
  Male- Pubic hair development- Week 52: Stage I | 1
  Male- Pubic hair development- Week 52: Stage II | 1
  Male- Pubic hair development- Week 52: Stage III | 2
  Male- Pubic hair development- Week 52: Stage IV | 6
  Male- Pubic hair development- Week 52: Stage V | 14
  Male- Pubic hair development- Week 156: number analyzed (Participants) | 14
  Male- Pubic hair development- Week 156: Stage I | 0
  Male- Pubic hair development- Week 156: Stage II | 0
  Male- Pubic hair development- Week 156: Stage III | 1
  Male- Pubic hair development- Week 156: Stage IV | 3
  Male- Pubic hair development- Week 156: Stage V | 10

80. Secondary Outcome: Change From Week 52 in Bone Age Assessment (X-ray of Left Hand and Wrist)- Week 156
Description: Change in bone age from week 52 to week 156. This outcome measure is applicable only for the Liraglutide 1.8 mg treatment arm.
Time Frame: Week 52, week 156
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Liraglutide 1.8 mg: Follow-up 1 and 2
Number analyzed (Participants) | 9
Years | 1.778 (1.277)

ADVERSE EVENTS:
Time Frame: Week 0 - 156. All presented AEs are TEAEs. A TEAE was defined as an event that had onset date on or after the first day of exposure to trial product and no later than 7 days after the last day of trial product administration.
Description: Adverse events were reported per reporting group for treatment period and follow up period. Results are based on SAS which included subjects: who received at least one dose of liraglutide or placebo for "Liraglutide 1.8 mg- Treatment period" and "Placebo" and who received liraglutide for more than 3 months during treatment period (week 0-52) and provided follow-up data anytime during weeks 53-104 for "Liraglutide 1.8 mg: Follow-up 1" and weeks 105-156 for "Liraglutide 1.8 mg: Follow-up 2".
Groups:
- Liraglutide 1.8 mg: Follow-up 2: Subjects who received liraglutide for more than 3 months during the treatment period (week 0-52), were followed-up at week 156.
Arm/Group | Liraglutide 1.8 mg | Placebo | Liraglutide 1.8 mg: Follow-up 1 | Liraglutide 1.8 mg: Follow-up 2
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/68 | 0/52 | 0/48
Serious Adverse Events (participants affected / at risk) | 9/66 | 4/68 | 7/52 | 2/48
Other Adverse Events (participants affected / at risk) | 45/66 | 49/68 | 7/52 | 1/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 1.8 mg (N=66) | Placebo (N=68) | Liraglutide 1.8 mg: Follow-up 1 (N=52) | Liraglutide 1.8 mg: Follow-up 2 (N=48)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fasciotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malocclusion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 1.8 mg (N=66) | Placebo (N=68) | Liraglutide 1.8 mg: Follow-up 1 (N=52) | Liraglutide 1.8 mg: Follow-up 2 (N=48)
Abdominal pain (Gastrointestinal disorders) | 11 (22) | 5 (6) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 8 (9) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 4 (5) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 15 (21) | 11 (13) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 8 (10) | 2 (4) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (10) | 6 (11) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 7 (8) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 14 (27) | 13 (39) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 4 (6) | 6 (9) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (16) | 19 (28) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 19 (25) | 9 (12) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 6 (10) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (5) | 4 (6) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (5) | 5 (5) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (4) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (10) | 5 (8) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 17 (46) | 6 (8) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT01541215/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT01541215/SAP_001.pdf